CLINICAL TRIAL: NCT01543776
Title: A Prospective Randomized Pilot Study Evaluating the Food Effect on the Pharmacokinetics and Pharmacodynamics of Abiraterone Acetate in Men With Castrate Resistant Prostate Cancer
Brief Title: Food Effect Study of Abiraterone Acetate for Treatment of Patients With Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0709; NCI-2012-00116 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-15; First posted 2012-03-05 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Castration-resistant Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (fasting) (Active Comparator): Patients receive abiraterone acetate PO daily first thing in morning after an overnight fast of at least 8 hours.
  Interventions: Drug: abiraterone acetate
- Arm II (fed) (Experimental): Patients receive abiraterone acetate PO daily within 30 minutes of a conventional low-fat breakfast.
  Interventions: Drug: abiraterone acetate

INTERVENTIONS:
Drug: abiraterone acetate — Given PO
  Other Names: CB7630; Zytiga

SUMMARY:
This randomized phase II trial studies the best way to give abiraterone acetate in treating patients with castration-resistant prostate cancer. Abiraterone acetate is effective in treating castrate resistant prostate cancer and is taken in the fasting state. However, the body's absorption of abiraterone is increased with food intake. This study will test the whether a lower dose of abiraterone taken with food has a similar effect on prostate specific antigen (PSA) compared to full dose taken fasting.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the pharmacodynamic effect of reduced dose (250mg daily) abiraterone acetate in the prandial state (250mg-Fed) to the full, standard 1000mg daily dose in the fasting state (1000mg-Fasting) as assessed by change in serum prostate-specific antigen (PSA).

SECONDARY OBJECTIVES:

I. To evaluate the effect of prandial states on plasma levels and the intra-patient pharmacokinetic variability of abiraterone acetate.

II. To evaluate the safety profile of reduced dose abiraterone acetate taken in the prandial state.

III. To evaluate the pharmacodynamic effect of reduced dose abiraterone acetate in the prandial state as assessed by reduction in the extra-gonadal androgen dihydroepiadrosterone sulfate (DHEA-S) and dihydroepiandrostenedione (DHEA).

IV. To evaluate the effect of prandial state on time to disease progression (Working group criteria).

OUTLINE: Patients are randomized to one of two treatment arms.

ARM I: Patients receive abiraterone acetate orally (PO) daily first thing in morning after an overnight fast of at least 8 hours.

ARM II: Patients receive abiraterone acetate PO daily within 30 minutes of a conventional low-fat breakfast.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Both arms will also be treated with prednisone 5mg twice daily.

After completion of study treatment, patients are followed up within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer with progressive disease defined as either:

  * 2 or more new lesions on bone scan or
  * Progressive disease on computed tomography (CT)/magnetic resonance imaging (MRI) according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria or
  * Rising prostate-specific antigen (PSA): PSA evidence for progressive prostate cancer consists of a minimum PSA level of at least 2 ng/ml, which has subsequently risen on at least 2 successive occasions, at least 2 weeks apart
* Evidence of castration resistance defined as disease progression despite a testosterone level < 50 ng/dL (or surgical castration)
* Any prior therapy for castrate disease is acceptable except prior abiraterone, which is excluded; a minimum washout of 28 days for any other anticancer therapy prior to first dose of study drug is required

  * Any other radiotherapy or radionuclide require 28-day washout prior to first dose of study drug
  * Denosumab or zoledronic acid are allowed
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Total bilirubin =< 1.5 x the upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Therapy with other hormonal therapy, including any dose of megestrol acetate (Megace), finasteride (Proscar), dutasteride (Avodart), or any herbal product known to decrease PSA levels (e.g., saw palmetto and PC-SPES), or any systemic corticosteroid (other than prednisone =< 10 mg/day) within 4 weeks prior to first dose of study drug
* Therapy with supplements or complementary medicines/botanicals within 4 weeks of first dose of study drug is excluded with the following exceptions:

  * Conventional multivitamin supplements
  * Selenium
  * Lycopene
  * Soy supplements
* Inability to swallow capsules or known gastrointestinal malabsorption
* History of other malignancies, with the exception of adequately treated non-melanoma skin cancer or adequately treated superficial bladder cancer or other solid tumors curatively treated with no evidence of disease for >= 5 years from enrollment
* Blood pressure that is not controlled despite > 2 oral agents (systolic blood pressure [SBP] > 160 and diastolic blood pressure [DBP] > 90 documented during the screening period with no subsequent blood pressure readings < 160/100)
* Serum potassium (K)+ < 3.5 mmoL/L on more than one reading within the screening period
* Serious intercurrent infections or non-malignant medical illnesses that are uncontrolled
* Active psychiatric illness/social situations that would limit compliance with protocol requirements
* New York Heart Association (NYHA) class II, NYHA class III, or IV congestive heart failure (any symptomatic heart failure)
* Concurrent therapy with strong inhibitors or inducers of Cytochrome P450 (CYP)3A4 due to concerning possible drug-drug interactions with abiraterone

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-01; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Szmulewitz, Principal Investigator — University of Chicago
Locations (6):
- United States (5):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - North Shore University Health System, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois Cancer Care, Peoria, Illinois
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Heiss BL, Geynisman DM, Martinez E, Wong ASC, Yong WP, Szmulewitz RZ, Stadler WM. Comparison of out-of-pocket costs and adherence between the two arms of the prospective, randomized abiraterone food effect trial. Support Care Cancer. 2022 Mar;30(3):2803-2810. doi: 10.1007/s00520-021-06670-3. Epub 2021 Nov 29. PMID 34845502
- [Derived] Szmulewitz RZ, Peer CJ, Ibraheem A, Martinez E, Kozloff MF, Carthon B, Harvey RD, Fishkin P, Yong WP, Chiong E, Nabhan C, Karrison T, Figg WD, Stadler WM, Ratain MJ. Prospective International Randomized Phase II Study of Low-Dose Abiraterone With Food Versus Standard Dose Abiraterone In Castration-Resistant Prostate Cancer. J Clin Oncol. 2018 May 10;36(14):1389-1395. doi: 10.1200/JCO.2017.76.4381. Epub 2018 Mar 28. PMID 29590007

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Fasting) | Arm II (Fed)
Started | 36 | 36
Completed | 34 | 34
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Fasting) | Arm II (Fed) | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Median (Full Range); unit: years] | 74 [54 to 82] | 72 [56 to 88] | 73 [54 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 36 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 17 | 43
  African American | 5 | 11 | 16
  Asian | 5 | 7 | 12
  Missing | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Singapore | 4 | 6 | 10
  United States | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in PSA Level
Description: Data were analyzed on a log scale: log(week 12) - log(baseline) = log ratio. Smaller (more negative) values indicate a better outcome.
Time Frame: From baseline to 12 weeks
Population: Two patients in each arm had missing data at 12 weeks.
Measure: Mean (Standard Error); unit: log ratio
Arm/Group | Arm I (Fasting) | Arm II (Fed)
Number analyzed (Participants) | 32 | 32
log ratio | -1.19 (0.29) | -1.59 (0.27)
Statistical Analysis 1: Comparison: Arm I (Fasting) vs Arm II (Fed); Test type: Non-Inferiority — The above criteria for non-inferiority corresponds to a response rate in the low dose arm that is no more than 15% lower than the response rate in the high dose arm (i.e., non-inferiority margin of 15%), under the assumption that the log ratios are approximately normally distributed; p < 0.10, t-test, 1 sided — Calculated p-value; Mean Difference (Final Values) = 0.3976, 90% CI 1-sided [lower limit -0.1111]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time to PSA progression (25% increase from baseline), radiographic progression, or death.
Time Frame: Assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Fasting) | Arm II (Fed)
Number analyzed (Participants) | 34 | 34
Months | 8.6 [3.6 to 11.0] | 8.6 [3.7 to 14.7]
Statistical Analysis 1: Comparison: Arm I (Fasting) vs Arm II (Fed); Test type: Superiority; p = 0.38, Log Rank

3. Secondary Outcome: Adrenal Androgen Production (DHEA-S)
Description: Extragonadal serum adrogen
Time Frame: Cycle 4 (4 months)
Population: 29 patients had missing data
Measure: Mean (Standard Error); unit: microgram per deciliter
Arm/Group | Arm I (Fasting) | Arm II (Fed)
Number analyzed (Participants) | 19 | 20
microgram per deciliter | 13.30 (1.47) | 10.22 (1.33)
Statistical Analysis 1: Comparison: Arm I (Fasting) vs Arm II (Fed); Test type: Superiority; p = 0.13, t-test, 2 sided

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Patients with grade 3 or higher AE (CTCAE Version 4.03)
Time Frame: Assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Fasting) | Arm II (Fed)
Number analyzed (Participants) | 34 | 34
Participants | 6 | 11
Statistical Analysis 1: Comparison: Arm I (Fasting) vs Arm II (Fed); Test type: Superiority; p = 0.26, Fisher Exact

5. Secondary Outcome: Peak Plasma Concentration of Abiraterone
Description: Analyzed on a log scale due to skewness of distribution
Time Frame: Up to 4 months
Population: Three patients had missing data.
Measure: Mean (Standard Error); unit: log(ng/mL)
Arm/Group | Arm I (Fasting) | Arm II (Fed)
Number analyzed (Participants) | 30 | 31
log(ng/mL) | 5.39 (0.19) | 4.65 (0.21)
Statistical Analysis 1: Comparison: Arm I (Fasting) vs Arm II (Fed); Test type: Superiority; p = 0.012, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm I (Fasting) | Arm II (Fed)
All-Cause Mortality (participants affected / at risk) | 6/34 | 4/34
Serious Adverse Events (participants affected / at risk) | 5/34 | 2/34
Other Adverse Events (participants affected / at risk) | 32/34 | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Fasting) (N=34) | Arm II (Fed) (N=34)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Fever (General disorders) | 1 | 0
General disorders and administrative site conditions (General disorders) | 1 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Infections and infestations-other (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Fasting) (N=34) | Arm II (Fed) (N=34)
Alanine aminotransferase increased (Investigations) | 4 | 2
Alkaline phosphatase increased (Investigations) | 3 | 2
Anemia (Blood and lymphatic system disorders) | 6 | 3
Anorexia (Metabolism and nutrition disorders) | 3 | 5
Anxiety (Psychiatric disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Constipation (General disorders) | 5 | 3
Depression (Psychiatric disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 5 | 4
Dizziness (Nervous system disorders) | 3 | 4
Dysphagia (Gastrointestinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Edema limbs (General disorders) | 5 | 4
Fatigue (General disorders) | 16 | 16
Fever (General disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 1
Hot flashes (Vascular disorders) | 6 | 2
Hypertension (Vascular disorders) | 10 | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 5
Hypokalemia (Metabolism and nutrition disorders) | 5 | 7
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Infections and infestations-Other (Infections and infestations) | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 3
Pain (General disorders) | 9 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5
Urinary frequency (Renal and urinary disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Chills (General disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Creatinine increased (Investigations) | 0 | 3
Eye disorders - Other (Eye disorders) | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Localized edema (General disorders) | 0 | 4
Musculoskeletal and connective tissue disorder-Other (Musculoskeletal and connective tissue disorders) | 0 | 4
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Platelet count decreased (Investigations) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3
White blood cell decreased (Investigations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT01543776/Prot_SAP_000.pdf